CLINICAL TRIAL: NCT04803409
Title: Ultrasound Neural and Immunomodulation Treatment Evaluation Study (UCSD-SW) for COVID-19
Brief Title: UNITE Study (UCSD-SW) for COVID-19
Acronym: UNITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imanuel Lerman (Other)
Collaborators: SecondWave Systems Inc. (Industry); MCDC (Unites States Department of Defense) (Unknown)
Responsible Party: Sponsor-Investigator, Imanuel Lerman, Asst Clin Prof, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201611
Record Dates: First submitted 2021-03-16; First posted 2021-03-17 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Intervention Model Description: The participants will be randomized to two groups: ultrasound group and control group. All participants will still receive standard clinical care. The ultrasound group will receive daily ultrasound application to the spleen for up to 7 days, in addition to the standard clinical care. The control group will receive standard clinical care without ultrasound stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Group (Experimental): Daily ultrasound application to the spleen of approximately 18 minutes for up to 7 days, in addition to standard clinical care.
  Interventions: Device: Splenic Ultrasound
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Device: Splenic Ultrasound — Splenic Ultrasound: Daily ultrasound application to the spleen of approximately 18 minutes for up to 7 days, in addition to standard clinical care
  Arms: Ultrasound Group

SUMMARY:
The research objective of the UNITE Study is to assess the potential efficacy of ultrasound application to the spleen using a small wearable ultrasound system in the treatment of coronavirus disease 2019 (COVID-19) in a pilot study.

Specific Aims:

Determine the efficacy of splenic ultrasound in affecting markers of systemic inflammation in COVID-19 infection.

Evaluate the potential efficacy of splenic ultrasound in affecting clinical outcomes in COVID-19 infection.

Condition or disease:

Covid19:

Cytokine Storm Inflammation

Device:

Splenic Ultrasound

Phase:

Not Applicable

DETAILED DESCRIPTION:
Detailed Description:

Ultrasound is widely used in human medicine because it is safe, non-invasive, and painless. The same kind of ultrasound that is used for imaging (for example, to visualize babies in utero) may be able to treat inflammatory diseases including COVID-19. COVID-19 is a disease caused by infection with the SARS-CoV-2 virus. Some COVID-19 patients develop a severe respiratory disease called acute respiratory distress syndrome and this disease is caused, in part, by a significant increase in inflammatory factors. Clinical therapies that reduce this elevated inflammation in the body (e.g., inflammation molecules in your body called cytokines) may be capable of diminishing symptoms in severe cases of COVID-19.

Multiple studies in animals with hyper-inflammation conditions (e.g., inflammatory arthritis and sepsis/LPS injections) and recent human studies (e.g., for the treatment of joint inflammation in Rheumatoid Arthritis) have shown that ultrasound applied to the spleen can suppress blood/genetic markers of inflammation. Similar inflammatory markers, or cytokines, are elevated in the lungs of COVID-19 patients and believed to cause severe symptoms. Splenic ultrasound can potentially lower these inflammatory cytokines without hindering antibody production, leading to clinical improvements in COVID-19 patients.

This study will employ investigational ultrasound devices produced by SecondWave Systems called the MINI System (Miniature Immunotherapy and Neuromodulation Instrument System).

There will be two groups in this study with 20 participants in each group. One group will receive ultrasound application to the spleen, in addition to the standard clinical care. A control group will receive standard clinical care without splenic ultrasound. Each ultrasound application session will last about 30 minutes per day for 7 days, unless the participant is discharged sooner. For ultrasound stimulation, a small wearable ultrasound device is positioned on the upper left abdomen area over the ribs. The ultrasound session on the first study day includes a period of 5-10 minutes when study personnel use an ultrasound imaging device to locate the spleen and to position the wearable MINI device in a proper location around the ribs area, and an approximately 18-minute period for application of ultrasound to the spleen. Collection of clinical outcome data and daily blood draws will be performed in each participant throughout the study through Day 8. Additional data collected from each participant during their routine clinical care beyond their study involvement will also be analyzed together with the study data to evaluate the specific aims of the clinical trial.

Study Design Go to sections Study Type : Interventional (Clinical Trial) Estimated Enrollment : 40 participants Allocation: Randomized Intervention Model: Parallel Assignment Intervention Model Description: The participants will be randomized to two groups: ultrasound group and control group. All participants will still receive standard clinical care. The ultrasound group will receive daily ultrasound application to the spleen for up to 7 days, in addition to the standard clinical care. The control group will receive standard clinical care without ultrasound stimulation.

Primary Purpose: Other

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Positive for SARS-CoV-2 (via PCR)
* Decreased blood oxygen saturation: Room air SaO2 < 94% and/or requiring supplemental oxygen at a flow rate of 2 L/min or greater.
* Admission to the hospital

Exclusion Criteria:

* Pregnant women
* Mechanically ventilated (if patient goes onto mechanical ventilation while participating in the study, they can continue ultrasound treatment if recommended by standard of care clinician and investigators of the study)
* Comfort care status
* On-duty Federal Employees and Military Personnel
* Patient without decision making capacity as determined by clinical judgement informed by communication with the UCSD primary Hospitalist team
* Any other clinical reasons deemed by the investigators of the study in which the patient would not be an appropriate candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
IL-6 Change | Baseline to Day 8 (end of treatment; or date of discharge)
  Between-arm change of IL-6 levels from baseline to end of treatment between groups
IL-1β | Baseline to Day 8 (end of treatment; or date of discharge
  Between-arm change of IL-1β levels from baseline to end of treatment between groups
CRP | Baseline to Day 8 (end of treatment; or date of discharge)
  Between-arm change of CRP levels from baseline to end of treatment between groups

SECONDARY OUTCOMES:
Change in time to recovery | Baseline to date of recovery, assessed up to 6 months
  Day of recovery is defined as the first day on which the subject satisfies this category from the ordinal scale: Hospitalized, no oxygen therapy

OTHER OUTCOMES:
Change in death rate | : Baseline to date of discharge or date of death, whichever came first, assessed up to 6 months
  Change in death rate
Change in rate of requiring mechanical ventilation | Baseline to date of discharge or date of death, whichever came first, assessed up to 6 months
  Change in rate of requiring mechanical ventilation
Change in duration of hypoxemia | Baseline to date of discharge or date of death, whichever came first, assessed up to 6 months
  Change in duration of hypoxemia
Change in serum cytokine concentration of TNF | Baseline to Day 8 (end of treatment; or date of discharge)
  Change in serum cytokine concentration of TNF
Change in serum cytokine concentration of IL-10 | Baseline to Day 8 (end of treatment; or date of discharge)
  Change in serum cytokine concentration of IL-10
Change in serum cytokine concentration of IFN-gamma | Baseline to Day 8 (end of treatment; or date of discharge)
  Change in serum cytokine concentration of IFN-gamma
Change in serum cytokine concentration of IL-18 | Baseline to Day 8 (end of treatment; or date of discharge)
  Change in serum cytokine concentration of IL-18
Change in serum cytokine concentration of IL2R-alpha | Baseline to Day 8 (end of treatment; or date of discharge)
  Change in serum cytokine concentration of IL2R-alpha
Change in serum cytokine concentration of IL-4 | Baseline to Day 8 (end of treatment; or date of discharge)
  Change in serum cytokine concentration of IL-4
Change in D-dimer levels | Baseline to Day 8 (end of treatment; or date of discharge
  Change in D-dimer levels

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No